CLINICAL TRIAL: NCT04397861
Title: T Cell Memory Fuels the Innate Response in Chronic CF Lung Disease
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SAAVED16GO
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to define the role of CD4+ and CD8+ T cell memory responses in the immunologic failure of patients with cystic fibrosis (CF) to clear infections. In a normal host, the immune system clears pathogens upon re-infection more swiftly and efficiently than during an initial infection, in great part due to the recall and effector functions of memory T cells. In CF, far less is understood regarding the response of T cell memory when hosts reencounter antigens, otherwise known as pulmonary exacerbations. Pulmonary exacerbations are pivotal events that lead to a decline in health status among CF patients, with many never recovering to baseline health. CF patients will be recruited from patients followed by the Adult CF Program at National Jewish Health. Following enrollment at the time of antibiotic initiation, blood will be collected at two different time points. The first samples will be collected within 24 hours of starting IV antibiotic therapy. The second blood specimen will be collected at the end of hospitalization, after a minimum of 5 days. At the time of each blood draw, complete blood counts, a sputum sample, and simple spirometry will be measured as part of the standard care of a CF exacerbation. Isolated PBMCs will be stained with antibodies to designate cell surface phenotype. They will then be sorted to identify the T cell population. These cells will be tested on their ability to clear pathogens. The relationship between cellular immune responses and clinical indicators of pulmonary status will be examined by fitting linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF.
* Age 18 years old or greater.
* Hospitalization with planned IV antibiotic treatment for a pulmonary exacerbation of CF.
* Ability to perform reproducible Pulmonary Function Tests and produce sputum.
* Willingness to comply with study procedure and willingness to provide written consent.

Exclusion Criteria:

* Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.
* Use of systemic steroids at the start of IV treatment for a pulmonary exacerbation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CF subjects will be recruited from patients followed by the Adult CF Program at National Jewish Health at the onset of an acute pulmonary exacerbation.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluate CD4+ and CD8+ T cell function during CF pulmonary exacerbation | average 10 days
  Prospectively evaluate CD4+ and CD8+ T cell function as measured from the peripheral blood in patients with cystic fibrosis (CF) and its correlation with improvements in pulmonary inflammation and clinical status during treatment of CF pulmonary exacerbations.
Evaluate CD4+ and CD8+ T cell function during CF pulmonary exacerbation | a period of 60 months
  Prospectively evaluate CD4+ and CD8+ T cell function as measured from the peripheral blood in patients with cystic fibrosis (CF) and its correlation with improvements in pulmonary inflammation and clinical status during treatment of CF pulmonary exacerbations.
Test the capacity of enhanced CFTR activity to bolster host inflammatory cell function | average 10 days
  Compare CF effector memory responses between those clinically prescribed a CFTR modulator and those not currently on treatment as measured by flow cytometry. The ability of CF effector T cells to control infection over time will change over the subject's lifetime and use of CFTR modulators.
Test the capacity of enhanced CFTR activity to bolster host inflammatory cell function | a period of 60 months
  Compare CF effector memory responses between those clinically prescribed a CFTR modulator and those not currently on treatment as measured by flow cytometry. The ability of CF effector T cells to control infection over time will change over the subject's lifetime and use of CFTR modulators.
Test the capacity of T cell subsets to control infection over time | average 10 days
  Compare CF effector memory responses between those who are infected frequently (2 or more times/year) and those infected infrequently (0-1 times/year) as measured by flow cytometry. The ability of CF effector T cells to control infection over time will change over the subject's lifetime and number of exacerbations.
Test the capacity of T cell subsets to control infection over time | a period of 60 months
  Compare CF effector memory responses between those who are infected frequently (2 or more times/year) and those infected infrequently (0-1 times/year) as measured by flow cytometry. The ability of CF effector T cells to control infection over time will change over the subject's lifetime and number of exacerbations.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No